CLINICAL TRIAL: NCT01167946
Title: Safety and Efficacy of Oral Mega Pulse Methylprednisolone in Severe Therapy Resistant Alopecia Areata
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: King Saud University (Other)
Collaborators: Saudi Society of Dermatology and Dermatologic surgery (Unknown)
Responsible Party: Ghada Binsaif, King Saud University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 03-451
Record Dates: First submitted 2010-07-21; First posted 2010-07-22 (Estimated); Last update posted 2010-07-22 (Estimated); Status verified 2003-01

CONDITIONS: Alopecia Totalis; Alopecia Universalis; Ophiasic Alopecia
Keywords: Alopecia Areata; Alopecia totalis; Alopecia Universalis; Ophiasic alopecia; Oral Pulse steroid; Methylprednisolone
MeSH Terms: conditions — Alopecia universalis; Alopecia Areata | interventions — Methylprednisolone Hemisuccinate

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group A (Experimental): will receive pulse treatment for 3 consecutive days once every 2 weeks for 24 weeks
  Interventions: Drug: methylprednisolone sodium succinate
- Group B (Active Comparator): will receive 2 consecutive daily pulses every 3 weeks for 24 weeks
  Interventions: Drug: methylprednisolone sodium succinate
- Group C (Active Comparator): will receive 3 consecutive daily pulses every 3 weeks for 24 weeks.
  Interventions: Drug: methylprednisolone sodium succinate

INTERVENTIONS:
Drug: methylprednisolone sodium succinate — Group A will receive pulse treatment for 3 consecutive days once every 2 weeks for 24 weeks. The daily dose of each pulse treatment will consist of methylprednisolone sodium succinate 15mg/kg of ideal body weight, given orally in 200 ml of fresh orange juice.
  Arms: Group A
Drug: methylprednisolone sodium succinate — Group B will receive 2 consecutive daily pulses every 3 weeks for 24 weeks. The daily dose of each pulse treatment will consist of methylprednisolone sodium succinate 15mg/kg of ideal body weight, given orally in 200 ml of fresh orange juice.
  Arms: Group B
Drug: methylprednisolone sodium succinate — Group C will receive 3 consecutive daily pulses every 3 weeks for 24 weeks. The daily dose of each pulse treatment will consist of methylprednisolone sodium succinate 15mg/kg of ideal body weight, given orally in 200 ml of fresh orange juice.
  Arms: Group C

SUMMARY:
Systemic Pulse Glucocorticoids have been shown to be effective in widespread Alopecia areata but not the totalis, universalis or ophiasic type. Whether the failure is due to inadequate dosing, inadequate frequency or other factors is a matter of debate. The investigators decided to conduct this study using the oral pulse steroid, however with higher doses and more frequent pulses to patients with severe forms of Alopecia areata.

DETAILED DESCRIPTION:
This will be a single-center, prospective, randomized study conducted in King Khalid University Hospital. Patients diagnosed with either Alopecia universalis, Alopecia totalis or Ophiasic alopecia will be included in the study. Patients with contraindications such as diabetes mellitus, peptic ulcer, hypertension, infection, psychosis, heart or kidney disease, endocrine disorders (apart from a subclinical hypothyroidism and autoimmune thyroiditis) will be excluded. Children less than 5 years of age and those who received systemic or topical treatment within the last 4 weeks before enrollment will be also excluded. Those of child bearing potential had to have a negative urine pregnancy test result at baseline visit and should practice a reliable method of contraception throughout the study. 42 eligible patients will be randomly assigned to one of 3 treatment groups. Enrolled patients must provide written informed consent. Institutional review board approval will be obtained.

ELIGIBILITY:
Inclusion Criteria:

* Alopecia Universalis
* Alopecia Totalis
* Ophiasic Alopecia

Exclusion Criteria:

* diabetes mellitus
* peptic ulcer
* hypertension
* infection
* psychosis
* heart disease
* kidney disease
* endocrine disorders (apart from a subclinical hypothyroidism and autoimmune thyroiditis)
* received systemic or topical treatment within the last 4 weeks before enrollment
* pregnancy

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2003-01; Primary Completion 2009-12 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
hair regrowth | at 36 weeks of treatment
  Photographs of scalp will be taken before treatment and every 2 visits. Analysis of the photographs will be conducted by two independent dermatologists. Primary efficacy measure will be the proportion of responders at 36 weeks.

SECONDARY OUTCOMES:
Safety of the protocol | from the first visit till one year after discontinuation of treatment
  Patients will be monitored for signs and symptoms of adverse events throughout study. Weight, temperature and blood pressure,Electrocardiography and serum electrolytes will be assessed at each visit. The followings will be also performed at specified time frame: complete blood count, blood biochemistry, electrocardiography, Chest x-ray, sinuses x-ray, Short synactin test, Bone mineral density and ophthalmologic examination.
Factors affect the response to treatment | at 36 weeks
  Responses will be analyzed in relation to clinical findings and presence of subclinical hypothyroidism, thyroid auto antibodies, antinuclear antibodies, ferritin level, IgE level and the presence and degree of dermal fibrosis, inflammation and epidermal follicular plugging

CONTACTS AND LOCATIONS:
Overall Officials: Ghada A Binsaif, MD, Principal Investigator — King Saud University
Locations (1):
- King Khalid University Hospital, Riyadh, Riyadh Region, Saudi Arabia